CLINICAL TRIAL: NCT05710263
Title: Bariatric Embolization Before Sleeve Gastrectomy for Super Obese Patients
Acronym: EMBOSLEEVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0043
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Sleeve Gastrectomy; Morbid Obesity; Bariatric Surgery
Keywords: bariatric embolization; sleeve gastrectomy; super obese; left gastric artery; Morbid Obesity; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: bariatric embolization — bariatric or left gastric artery embolization

SUMMARY:
In patients with severe obesity, bariatric surgery provides consistent and long-term weight loss. BMI ≥50kg / m2 is an independent factor of increased morbidity / mortality in bariatric surgery compared with patients weighing less than 50 kg / m2 (1.2% and 0.8%) mainly due to technical difficulties. Preoperative weight loss reduces this morbidity / mortality. Recent studies have shown that blocking blood vessels to a particular portion of the stomach (bariatric or left gastric artery embolization) can temporarily decrease levels of the appetite inducing hormone ghrelin, and result in weight loss. The purpose of this study was to evaluate the safety and effectiveness of the association bariatric embolization before sleeve gastrectomy in super obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing, able and mentally competent to provide written informed consent.
* Body mass index (BMI) >50kg/m².
* 3 risk factors (De Maria et al) among: hypertension, male gender, age>45, risk of pulmonary embolism
* Vascular anatomy (including celiac, hepatic, and gastric arteries) that in the opinion of the interventional radiologist amenable to Bariatric Embolization, as assessed on 3D CT angiography.
* Adequate hematological, hepatic and renal function as follows:

Hematological Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L INR <1.5 Hepatic Bilirubin ≤ 2.0 mg/dL Albumin ≥ 2.5 g/L Renal Estimated GFR > 60ml/min.1.73m2

* Aged 18 years or older.
* Patient who is going to be operated by sleeve gastrectomy

Exclusion Criteria:

* Prior history of gastric pancreatic, hepatic, and/or splenic surgery
* Prior radiation to the upper abdomen
* Prior embolization to the stomach, spleen or liver
* Portal venous hypertension
* Prior or current history of peptic ulcer disease
* Significant risk factors for peptic ulcer disease including daily NSAID use and smoking.
* Active H. Pylori infection
* Weight greater than 240 kg
* Known aortic pathology such as aneurysm or dissection renal insufficiency as evidenced by an estimated glomerular filtration rate of < 60 milliliters per minute
* Major comorbidity such as cancer, significant cardiovascular disease, diabetes, or peripheral arterial disease.

Pregnancy

* ASA Class 4 or 5 (very high risk surgical candidates: class 4= incapacitating disease that is a constant threat to life) at the time of screening for enrollment into the study will be excluded from participation. This exclusion criterion exists because of the possibility that surgical intervention will be needed if the study intervention subsequently leads to severe adverse effects.
* History of Inflammatory Bowel Disease
* Cirrhosis
* Known history of allergy to iodinated contrast media
* Contraindications to use Embosphere (ex:known allergy to gelatin ..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
NUmber of Adverse Events | 12 months

SECONDARY OUTCOMES:
Weight Loss | 12 months
  Unit of Measure: Percentage of excess weight loss

IPD SHARING:
Plan to Share IPD: No